CLINICAL TRIAL: NCT07095374
Title: Associations Between Radiographic Inclination of Premolars and Maxillary Expansion: Retrospective Observational Study
Brief Title: Associations Between Radiographic Inclination of Premolars and Maxillary Expansion
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Other Study IDs: 2025-PREMOLARSEXPANSION
Record Dates: First submitted 2025-06-26; First posted 2025-07-31 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Maxillary Deficiency
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthodontic patients undergone rapid palatal expander treatment: Patients treated with rapid palatal expansion. Patients must have a pre-treatment and post-treatment orthopantomography.
  Interventions: Other: Rapid palatal expansion

INTERVENTIONS:
Other: Rapid palatal expansion — Patients undergone orthopedic treatment with rapid palatal expander

SUMMARY:
Recruitment of patients treated using rapid maxillary expanders with dental anchorage, with pre-treatment panoramic X-rays and post-treatment models. In the initial phase of the study, the objective is to correlate the radiographic inclination of the upper permanent premolars in the pre-treatment orthopantomography to the expansion obtained at the end of therapy using a palatal expander with dental anchorage.

DETAILED DESCRIPTION:
Maxillary transverse deficiency is a common malocclusion, frequently associated with unilateral or bilateral posterior crossbite, with a prevalence ranging from 8% to 22%. Since transverse development occurs earlier than vertical and sagittal development, inadequate transverse growth can also affect overall craniofacial development. This deficiency can impact aesthetics and functions such as creating excessive buccal corridor spaces, causing dental crowding, and reducing nasal cavity volume, which can lead to breathing difficulties. Thus, timely correction of maxillary transverse deficiency is crucial for harmonizing the relationship between the upper and lower jaws, as well as for enhancing aesthetics and functionality. Currently, rapid maxillary expansion (RME) is a widely accepted and established treatment for correcting maxillary constriction in patients during their peak growth period.

There is no protocol in the literature that investigates the need for transverse expansion of the upper jaw through the analysis of the inclination of the long axis of the upper premolars and canines. Therefore, the aim of this study is to investigate the predictability of the necessary expansion through the analysis of the inclination of the upper premolars and canines in orthopantomography.

In this retrospective study, patients who are scheduled for treatment using rapid palatal expanders with dental anchorage will be recruited. A requirement for recruitment will be the presence of pre-treatment orthopantomography.

The inclination of the tooth will be calculated between the long axis of the tooth and the middle line as previously described by Baccetti et all. In their works regarding impacted canines.

The achieved expansion will be evaluated based on the number of activations recorded in each individual patient's chart clinical records.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for orthopedic treatment with rapid palatal expander
* Pre-treatment orthopantomography
* Pre and post treatment intraoral scan

Exclusion Criteria:

* Previous maxillofacial surgery
* cleft lip and palate
* premolar agenesis or extraction for fracture ecc.
* Previous orthopedic-orthodontic treatments

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients referring to the Unit of Orthodontics and Pediatric Dentistry for oral care
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of required activation for maxillary expansion | T0 (pre-treatment casts/x-rays) and T1 (post-treatment casts/x-rays)
  Correlation between the number of activations of the rapid palatal expander and premolar inclination (angle between the long axis of the premolars with the occlusal plane)

SECONDARY OUTCOMES:
Canine inclination | T0 (pre-treatment x-rays) and T1 (post-treatment x-rays)
  Angle between canines and the occlusal plane

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, phD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the principal investigator.